CLINICAL TRIAL: NCT06386718
Title: Comparison of Ultrasonographic Measurements of Radial and Ulnar Arteries in Pediatric Patients Undergoing Elective Surgery
Brief Title: Ultrasonographic Evaluation of Arteries of the Hand in Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ozlem Can, Professor, Ankara University
Other Study IDs: USG for ped art can
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Ulnar and Radial Artery
Keywords: ultrasonography for cannulation; pediatrics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasound measurements of the ulnar artery and radial artery at different angles are obtained and compared to determine the optimal diameters for possible arterial cannulation in pediatric patients.

DETAILED DESCRIPTION:
Radial artery cannulation is the most commonly used technique for invasive arterial catheterization in pediatric patients. Ultrasound guidance has significantly reduced cannulation success rates and complication risks. The ulnar artery presents an anatomical alternative to the radial artery and has emerged as a potential cannulation site. This study aims to comprehensively evaluate the suitability of the radial or ulnar artery for cannulation in pediatric patients.

Finding of this study objectives are

To obtain a large sample of pediatric patients from different age groups To measure arterial diameters using ultrasound at different angles and with ultrasound and to assess the optimal artery and the angle.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 or 2
* Patients scheduled for elective surgical procedures
* Informed consent must be obtained from both the patient and, if applicable, their parent or guardian.

Exclusion Criteria:

* Patients over 10 years of age
* Patients with congenital anomalies or syndromic conditions
* Abnormal Allen Test
* Skin Erosion or infection at the cannulation site
* Hematoma at the cannulation site

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Between 0 and 10 years of ages pediatric patients scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determining the Diameter and Depth at different angles | only once
  The study aims to measure the radial and ulnar arteries using ultrasound at different angles to determine the widest diameter and the optimal angle to achieve this diameter.
Comparing Ulnar and Radial Artery Diameters Across Age Groups | only once
  Investigating whether there is a difference (ulnar>radial, ulnar=radial, or radial>ulnar) in the diameter of the ulnar artery compared to the radial artery among the age groups included in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Ankara, Turkey (Türkiye)